CLINICAL TRIAL: NCT07181447
Title: Quantitative Assessment of Pelvic Floor Muscle Fitness in Myofascial Pelvic Pain
Brief Title: NIRS for the Diagnosis of Myofascial Pelvic Pain
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Anne Lenore Ackerman, Associate Professor of Urology, University of California, Los Angeles
Other Study IDs: 22-0428; R61AT013008-01 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Myofascial Pelvic Pain
Keywords: pelvic pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control Subjects: Women age 18 or older without pelvic pain or other genitourinary complaints
  Interventions: Diagnostic Test: Pelvic Floor Muscle Assessment by Near-Infrared Spectroscopy
- Myofascial Pelvic Pain Subjects: Women age 18 or older with pelvic floor muscle pain or tender points
  Interventions: Diagnostic Test: Pelvic Floor Muscle Assessment by Near-Infrared Spectroscopy

INTERVENTIONS:
Diagnostic Test: Pelvic Floor Muscle Assessment by Near-Infrared Spectroscopy — This study will develop and test an instrument to establish a normal range for near infrared spectroscopy (NIRS) optical changes associate with pelvic floor exercise in adult women based on the test-to test (intra-day) reliability of oxygen kinetics related to contraction of the pelvic floor muscle. We will establish the relationship between the quantitative NIRS data, the condition of Myofascial pelvic musculature and the symptomatology of MPP and related comorbidities. We will also evaluate prospectively the effectiveness of these data in predicting effective treatment modalities. Finally, we will optimize a training regime for non-specialists to allow this technique to be used in a variety of settings. The development of this device and validation of its relevance to diagnosis and treatment of MPP will provide effective care sooner and at a lower cost than current procedures. It will also reduce inequities in the availability of care to underserved populations.

SUMMARY:
Myofascial Pelvic Pain (MPP) is an often-misdiagnosed condition affecting up to 26% of women during their lives and imposing enormous costs on national health care systems. It frequently involves comorbidities such as bladder, bowel, and sexual dysfunction. There are no quantitative measures that adequately guide the physician and accurate diagnosis typically requires an internal examination by a tertiary specialist.

This study will develop and test an instrument to establish a normal range for near infrared spectroscopy (NIRS) optical changes associate with pelvic floor exercise in adult women based on the test-to test (intra-day) reliability of oxygen kinetics related to contraction of the pelvic floor muscle.

We will establish the relationship between the quantitative NIRS data, the condition of Myofascial pelvic musculature and the symptomatology of MPP and related comorbidities. We will also evaluate prospectively the effectiveness of these data in predicting effective treatment modalities. Finally, we will optimize a training regime for non-specialists to allow this technique to be used in a variety of settings.

The development of this device and validation of its relevance to diagnosis and treatment of MPP will provide effective care sooner and at a lower cost than current procedures. It will also reduce inequities in the availability of care to underserved populations by providing an inexpensive, reliable and easily available method for a variety of providers to address MPP.

DETAILED DESCRIPTION:
DETAILED DESCRIPTION Introduction. Myofascial pelvic pain (MPP) is the predominant underlying cause in 60-90% of women with chronic pelvic pain. MPP can be debilitating, and is often associated with bladder, bowel, and sexual dysfunction. MPP can be debilitating, leading to social withdrawal, loss of productivity, impaired relationships, and psychological comorbidities. Despite the high prevalence, myofascial pain is often overlooked by first-line healthcare providers; most providers, including gynecologic and urologic specialists, lack the knowledge or experience to even identify MPP. Unfortunately, there are currently no widely accepted measures to quantify muscular fitness or dynamic function of the pelvic floor. Improved recognition of MPP needs objective, reproducible, and quantifiable assessments of PFM fitness, to differentiate between forms of myofascial dysfunction and correlate those patterns with different symptoms. Improved recognition of MPP needs objective, reproducible, and quantifiable assessments of PFM fitness, to facilitate improvements in the recognition and diagnosis of MPP.

Objective: This trial will use optical technology (near infrared spectroscopy) to provide novel imaging and physiologic measures relevant to the PFM for the diagnostic evaluation of MPP.

Subject Recruitment: Healthy controls, who must lack pelvic pain, bowel disturbances, urinary symptoms, or sexual dysfunction, will be recruited from the community through online and targeted advertisements in gynecology and primary clinics. IRB approval for these studies is already in place, and we have already begun recruitment of control volunteers. Subjects with MPP, defined by pelvic floor myofascial pain in the absence of other identifiable pain generators, will be recruited from the UCLA Center for Women's Pelvic Health.24 MPP subjects meeting inclusion/exclusion criteria will be approached for enrollment prior to treatment assignment. Baseline demographics and clinical data, including age, height, weight, comorbidities, past surgeries, and medications, including hormones, will be self-reported at enrollment through a questionnaire on REDCap.

Vaginal NIRS-based Pelvic Floor Assessment: An 8-channel, multipoint vaginal NIRS interface miniaturized into a tampon-sized instrument, capable of measuring regional changes in pelvic floor muscle oxygenation in different quadrants and muscle depths, will assess oxygenation and hemodynamic parameters in the pelvic floor muscles. The NIRS sensor, housed in a sterile, single use, disposable child size speculum and placed within a sterile cover, will be inserted in the vagina. The participant will then complete two rounds of the same standardized series of contractions: a series of three maximal voluntary contractions (MVC) and one sustained contraction (SMVC). After each contraction series, there will be a 2-minute recovery period.

Statistical Analysis. Individual NIRS parameters for MPP subjects will be compared to controls by independent sample t-test or Wilcoxon signed-rank test. To generate a predictive model for MPP diagnosis, we will use Least Angle Shrinkage and Selection Operator (LASSO) to identify candidate predictors from individual NIRS features using ten-fold cross-validation. From potential predictors (i.e., non-zero coefficients), we will select features with standardized shrunken coefficients >0.4 to be used in a multivariable logistic regression model. Only statistically significant model coefficients will be retained to provide a reduced predictive model, whose performance will be evaluated by area under the receiver operating curve (AUROC). AUROC values >0.7 will be demonstrative of an acceptable diagnostic test. We will also report the sensitivity, specificity, and accuracy of the model to quantify anticipated impact.

Outcome: NIRS-based algorithm for the diagnosis of MPP. Impact: The R61 phase will validate vaginal NIRS as an effective, non-invasive, and scalable method to assess pelvic floor muscle fitness, correlating well with current measures of PFM strength and distinguishing the myofascial dysfunction associated with MPP from healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 100 years of age
* Pelvic pain for more than 6 months duration
* Report an average daily pain intensity score of at least 4 (on a 0 to 10 scale)
* Palpable trigger/tender points in internal pelvic floor muscles on standardized myofascial pelvic floor exam
* Willing to refrain from new clinical treatments that may affect pain during the study period

Exclusion Criteria:

* Inability to participate in clinic visits
* Prior invasive pelvic procedures for pain (e.g., prior pelvic surgery, sacral neuromodulation, intradetrusor Botox®)
* Active UTI or vaginal infection
* Pregnancy, childbirth during the previous 12 months, currently planning pregnancy
* Illicit Drug addiction/regular use of controlled substances
* Malignancy or other serious medical condition (e.g., poorly controlled diabetes [HgA1c > 8], neurologic or rheumatic disease)
* Diagnosed with an alternate cause of pelvic pain (e.g., interstitial cystitis, vestibulodynia, vulvar dermatoses dysmenorrhea)
* Urinary retention
* Greater than stage 3 pelvic organ prolapse
* Indwelling vaginal devices (e.g., pessary, contraceptive ring)
* Inability to sign an informed consent, fill out questionnaires, or complete study interviews

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control subjects (cohort 1) will be adult 18 (>18 years of age) who lack pelvic pain or other genitourinary symptoms. The MPP cohort (cohort 2) will consist of adult women >18 years of age with pelvic floor muscle pain or tender points.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
MPP Diagnosis | 1 day
  Accurate Diagnosis of Myofascial Pelvic Pain

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center for Women's Pelvic Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed, deidentified data will be submitted to a generalist repository that is supported by the BioMedical Informatics Coordinating Committee (BMIC) of the NIH, specifically the Harvard Dataverse open-source research data repository (https://dataverse.org).
Supporting Information: Study Protocol, Analytic Code
Time Frame: After completion of the study, metadata will be shared for a minimum of five years.
Access Criteria: Deidentified data will be freely available.